CLINICAL TRIAL: NCT02410655
Title: An Evidence Based Protocol for Oxytocin Administration in Vaginal Delivery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Submission discarded. Study never enrolled subjects.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-00279; NCT02453568 (obsolete NCT alias)
Record Dates: First submitted 2015-04-02; First posted 2015-04-07 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Uterine Atony; Postpartum Hemorrhage
Keywords: Uterine atony; Postpartum hemorrhage; Vaginal delivery; Uterotonic; Oxytocin; Bolus; Evidence-based; Protocol
MeSH Terms: conditions — Uterine Inertia; Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional standard of care (Active Comparator): Traditional administration of oxytocin at Lutheran Medical Center involves the use of two 20 IU / 1000 mL bags hung sequentially at a flow rate of 125 mL / hour each after the delivery of the anterior shoulder. This will total no more than 16 hours.
  Interventions: Drug: Oxytocin
- Evidence based protocol (Active Comparator): The proposed evidence based protocol involves utilizing a single 30IU / 500mL bag of oxytocin. After the delivery of the anterior shoulder, an initial rapid infusion bolus of 50mL of the 30IU / 500mL at 999mL / hour. Three minutes after rapid infusion, uterine tone should be assessed. If inadequate uterine tone persists, a second rapid infusion at the same dose and rate as above should be given. If inadequate uterine tone persists, a third rapid infusion may be given. If adequate uterine tone is achieved after any rapid infusion, the remainder of the bag should be administered at a rate of 100mL / hour until finished. If adequate tone is not achieved, the remainder of the bag should be administered at 100mL / hour and additional uterotonic agents should be considered.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — 500 mL bag of oxytocin (30 IU / 500 mL) to be connected to the IV, and controlled at the obstetricians request. Up to two, 50 mL rapid infusion boluses to be given after delivery of anterior shoulder. Upon completing the bolus(es) flow rate should be continued at 100 mL / hour. This should total no more than 4.5 hours.
  Other Names: Pitocin
  Arms: Evidence based protocol
Drug: Oxytocin — A total of two 1000 mL bags of oxytocin (20 IU/ 1000 mL) are to be connected to the IV sequentially, and controlled at the obstetricians request, are each to be administered over 8 hours after delivery of anterior shoulder in vaginal delivery. This will total 16 hours of oxytocin infusion.
  Other Names: Pitocin
  Arms: Conventional standard of care

SUMMARY:
The purpose of this study will be to evaluate a standardized, evidence-based protocol versus a conventional approach for the dosing of oxytocin in vaginal delivery.

DETAILED DESCRIPTION:
A traditional practice in many US hospitals includes use of 10-40 IU of Oxytocin mixed in various volumes of crystalloid administered at an unspecified and uncontrolled rate (quite often off the pump) in order to restore uterine tone and minimize routine blood loss in the third stage of labor. Many practitioners question high dose oxytocin regimens, timing and duration of Oxytocin administration for postpartum hemorrhage prophylaxis. Given the lack of a universally accepted, evidence based protocol, this study aims at comparing the efficacy of a traditional approach of administration of Oxytocin with an evidence-based designed algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal Delivery

Exclusion Criteria:

* Cesarean Delivery
* Allergy to Oxytocin
* Cardiac Arrhythmia

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

PRIMARY OUTCOMES:
Estimated blood loss | 24 hours postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Violetta Lozovyy, MD, Principal Investigator — Lutheran Medical Center; Jade King, BS, Principal Investigator — Lutheran Medical Center; Roulhac D Toledano, MD, PhD, Study Director — Lutheran Medical Center; Kevin Fitzpatrick, MD, Study Chair — Lutheran Medical Center